CLINICAL TRIAL: NCT01934556
Title: A Phase I/II, Open Label, Multicenter, Randomized, Controlled Study of the Safety, Tolerability and Efficacy of Intravitreal Injections of 0.3 mg Ranibizumab Given Monthly Compared to a TReat and EXtend Protocol in Patients With Diabetic Macular Edema
Brief Title: A Safety and Efficacy Trial of a Treat and Extend Protocol Using Ranibizumab With and Without Laser Photocoagulation for Diabetic Macular Edema
Acronym: TREX-DME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Palmetto Retina Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ML28724
Record Dates: First submitted 2013-08-28; First posted 2013-09-04 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab; Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Monthly (Active Comparator): Monthly Cohort (30 eyes) - Study eyes will receive intravitreal injections of 0.3 mg ranibizumab every 4 weeks for 24 months.
  Interventions: Drug: Ranibizumab 0.3 mg intravitreal injection
- TREX (Active Comparator): (60 eyes) - Monthly intravitreal injections of 0.3 mg ranibizumab for four visits. At the fourth visit (Week 12), if the central foveal thickness is ≤ 325 μm then the eye will receive 0.3 mg ranibizumab and begin the extension phase of the study. For all subsequent visits in the extension phase, appropriate changes to the treatment interval with 0.3 mg ranibizumab (i.e. extend, maintain, reduce) will be made based on pre-specified SD (Spectral Domain)-OCT criteria. Treatment is rendered at every visit. The time between visits is individualized based on each subject's response to treatment. If the central foveal thickness is > 325 μm at week 12, then the patient will continue to receive monthly intravitreal injections of 0.3 mg ranibizumab until the central foveal thickness is ≤ 325 μm. Once the central foveal thickness is ≤ 325 μm, then the study eye will begin the extension phase of the study.
  Interventions: Drug: Ranibizumab 0.3 mg intravitreal injection
- GILA (Active Comparator): (60 eyes) - Monthly intravitreal injections of 0.3 mg ranibizumab for four visits combined with guided laser photocoagulation to all microaneurysms in the area of DME at visit 2 (Week 4) and then again every 3 months, if leakage is present on fluorescein angiography. If the central foveal thickness is ≤ 325 μm at visit 4 (Week 12), eyes will receive 0.3 mg ranibizumab and the extension phase will begin. For all subsequent visits in the extension phase, appropriate changes to the treatment interval with 0.3 mg ranibizumab (i.e. extend, maintain, reduce) will be made based on pre-specified SD-Optical coherence tomography criteria. If the central foveal thickness is > 325 μm at week 12, then the patient will continue to receive monthly intravitreal injections of 0.3 mg ranibizumab and possible guided laser every 3 months until the central foveal thickness is ≤ 325 μm. Once the central foveal thickness is ≤ 325 μm, then the study eye will begin the extension phase of the study.
  Interventions: Drug: Ranibizumab 0.3 mg intravitreal injection; Device: Guided Laser Photocoagulation

INTERVENTIONS:
Drug: Ranibizumab 0.3 mg intravitreal injection
  Other Names: Ranibizumab; Lucentis
Device: Guided Laser Photocoagulation
  Other Names: NAVILAS Guided Laser System
  Arms: GILA

SUMMARY:
The purpose of this research study is to determine if a "Treat and Extend" regimen (increasing the time between visits when the disease is stable and not getting worse) of Ranibizumab 0.3 mg injections inside the eye is safe and effective at treating patients with swelling of the retina from diabetes.

DETAILED DESCRIPTION:
This research study will compare the visual outcomes between a group of patients who are treated with monthly injections of Ranibizumab 0.3 mg and two groups of patients who are treated with the "Treat and Extend" regimen. One of the "Treat and Extend" groups will also receive laser therapy to determine if this has any additional beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years of age Patient related considerations
* For sexually active women of childbearing potential, agreement to the use of an appropriate form of contraception (or abstinence) for the duration of the study
* Although no birth control method is 100% effective, the following are considered effective means of contraception: surgical sterilization, use of oral contraceptives, barrier contraception using either a condom or diaphragm with spermicidal gel, an intrauterine device, or contraceptive hormone implant or patch. A patient's primary care physician, obstetrician, or gynecologist should be consulted regarding an appropriate form of birth control.
* Ability and willingness to return for all scheduled visits and assessments

Disease related considerations

* The presence of center-involving diabetic macular edema on clinical exam and SDOCT
* Best corrected visual acuity in the study eye, using ETDRS testing, between 20/25 and 20/320 (Snellen equivalent), inclusive.
* Clear ocular media and adequate pupillary dilation to permit good quality fundus imaging.

Exclusion Criteria:

* General Exclusion Criteria

  * Pregnancy (positive urine pregnancy test) or lactation.
  * Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD (Intrauterine Device) , or contraceptive hormone implant or patch.
  * Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
  * Participation in another simultaneous medical investigation or trial

Ocular Exclusion Criteria Prior Ocular Treatment

* History of active proliferative diabetic retinopathy in the study eye on clinical exam
* History of vitrectomy surgery, submacular surgery, or other intraocular surgical intervention for diabetic macular edema in the study eye
* Any previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection, anti-VEGF drugs including ranibizumab, or device implantation) in the study eye within 90 days of the screening visit.
* History of prior laser macular photocoagulation more than 90 days prior to screening will be eligible for study inclusion. However, if the investigator does not feel that additional laser photocoagulation can be safely performed or would benefit the patient, then the eye in consideration will be excluded.
* Evidence of vitreomacular interface abnormality or epiretinal membranes which may be responsible for macular edema

Concurrent Ocular Conditions

• Any concurrent intraocular condition in the study eye (e.g., cataract or macular degeneration) that, in the opinion of the investigator, could either: Require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition; or if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA (Best Corrected Visual Acuity) over the 24-month study period.

* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Intraocular surgery (including cataract surgery) in the study eye within 3 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as IOP (Intraocular Pressure) ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma-filtering surgery in the study eye
* History of corneal transplant in the study eye
* History of pars plana vitrectomy

Concurrent Systemic Conditions

* Any history of use of systemic anti-VEGF (Vascular Endothelial Growth Factor) agents
* Uncontrolled blood pressure (defined as systolic > 180 mmHg and/or diastolic > 110 mmHg while patient is sitting) If a patient's initial reading exceeds these values, a second reading may be taken 30 or more minutes later. If the patient's blood pressure needs to be controlled by antihypertensive medication, the patient can become eligible if medication is taken continuously for at least 30 days prior to Day 0.
* Atrial fibrillation not managed by patient's primary care physician or cardiologist within 3 months of screening visit
* Women of childbearing potential not using adequate contraception (as defined in the inclusion criteria).

A woman is considered not to be of childbearing potential if she is postmenopausal, defined by amenorrhea for at least 1 year in a woman > 45 years old; or has undergone hysterectomy and/or bilateral oophorectomy.

* History of stroke within the last 3 months of screening visit
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications
* Current treatment for active systemic infection
* Active malignancy
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the reading center
* Inability to comply with study or follow-up procedures
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Palmetto Retina Center, West Columbia, South Carolina
  - Retina Consultants of Houston, Houston, Texas

REFERENCES:
- [Derived] Payne JF, Wykoff CC, Clark WL, Bruce BB, Boyer DS, Brown DM; TREX-DME Study Group. Long-term outcomes of treat-and-extend ranibizumab with and without navigated laser for diabetic macular oedema: TREX-DME 3-year results. Br J Ophthalmol. 2021 Feb;105(2):253-257. doi: 10.1136/bjophthalmol-2020-316176. Epub 2020 Apr 17. PMID 32303499
- [Derived] Payne JF, Clark WL, Bruce BB, Wykoff CC, Brown DM, Menke BM, Iverson SM, Allen KF, Boyer DS; Treat & Extend Protocol in Patients with Diabetic Macular Edema Study Group. Retinopathy Regression with Treat and Extend Ranibizumab for Diabetic Macular Edema. Ophthalmology. 2018 Aug;125(8):1304-1306. doi: 10.1016/j.ophtha.2018.03.046. Epub 2018 May 3. No abstract available. PMID 29729809
- [Derived] Payne JF, Wykoff CC, Clark WL, Bruce BB, Boyer DS, Brown DM; TREX-DME Study Group. Randomized Trial of Treat and Extend Ranibizumab with and without Navigated Laser for Diabetic Macular Edema: TREX-DME 1 Year Outcomes. Ophthalmology. 2017 Jan;124(1):74-81. doi: 10.1016/j.ophtha.2016.09.021. Epub 2016 Nov 8. PMID 27836430

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Units are Eyes
Groups:
- TREX: (60 eyes) - Monthly intravitreal injections of 0.3 mg ranibizumab for four visits and then underwent a treat and extend protocol of ranibizumab without navigated laser therapy.
- GILA: (60 eyes) - Monthly intravitreal injections of 0.3 mg ranibizumab for four visits and then underwent a treat and extend protocol of ranibizumab with navigated laser therapy.
Period: Overall Study
Arm/Group | Monthly | TREX | GILA
Started | 30; 30 Units are Eyes | 60; 60 Units are Eyes | 60; 60 Units are Eyes
Completed | 25; 25 Units are Eyes | 44; 44 Units are Eyes | 50; 50 Units are Eyes
Not Completed | 5; 5 Units are Eyes | 16; 16 Units are Eyes | 10; 10 Units are Eyes
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 4 | 10 | 7
Not completed — Death | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Monthly: Monthly Cohort (30 eyes) - Study eyes will receive intravitreal injections of 0.3 mg ranibizumab every 4 weeks for 24 months.
  Ranibizumab 0.3 mg intravitreal injection
- TREX: (60 eyes) - Monthly intravitreal injections of 0.3 mg ranibizumab for four visits. At the fourth visit (Week 12), if the central foveal thickness is ≤ 325 μm then the eye will receive 0.3 mg ranibizumab and begin the extension phase of the study. For all subsequent visits in the extension phase, appropriate changes to the treatment interval with 0.3 mg ranibizumab (i.e. extend, maintain, reduce) will be made based on pre-specified SD (Spectral Domain)-OCT criteria. Treatment is rendered at every visit. The time between visits is individualized based on each subject's response to treatment. If the central foveal thickness is > 325 μm at week 12, then the patient will continue to receive monthly intravitreal injections of 0.3 mg ranibizumab until the central foveal thickness is ≤ 325 μm. Once the central foveal thickness is ≤ 325 μm, then the study eye will begin the extension phase of the study.
  Ranibizumab 0.3 mg intravitreal injection
- Total: Total of all reporting groups
Arm/Group | Monthly | TREX | GILA | Total
Number analyzed (Participants) | 30 | 60 | 60 | 150
Number analyzed (Eyes) | 30 | 60 | 60 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 58.7 [52.5 to 66.0] | 59.4 [54.2 to 65.2] | 59.9 [53.3 to 66.7] | 59.5 [53.5 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 32 | 24 | 72
  Male | 14 | 28 | 36 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 21 | 18 | 51
  White | 12 | 31 | 31 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 30 | 60 | 60 | 150
Body-Mass Index [Median (Inter-Quartile Range); unit: Units of measure "kg/m^2"] | 32.2 [29.0 to 33.7] | 31.9 [28.3 to 35.4] | 30.9 [27.5 to 35.3] | 31.6 [28.1 to 35.0]
Mean Duration of Diabetes [Mean (Inter-Quartile Range); unit: Years] | 15 [9.25 to 20] | 13.5 [9 to 19.25] | 13.5 [9 to 19.25] | 14 [9 to 19.25]
Phakic Status [Number; unit: participants] | 23 | 48 | 46 | 117
Mean Best Corrected Visual Acuity (ETDRS Letters) [Mean (Inter-Quartile Range); unit: units on a scale] — Best Corrected Visual Acuity (BCVA) was measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters. More letters read correctly results in a higher letter score, which represents better visual acuity
  units on a scale | 67.5 [55.3 to 72.8] | 65.5 [55.0 to 80.0] | 67.0 [59.8 to 73.0] | 66.5 [57.0 to 75.8]
Central Retinal Thickness (microns) [Number; unit: Microns] — The Central Retinal Thickness is measured using an OCT machine which scans the retina. The Lower number of microns is better
  Microns | 415 | 452 | 484 | 452

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Vision at 24 Months
Description: Mean change in ETDRS (Early Treatment in Diabetic Retinopathy Study) visual acuity at 24 months (week 92-week 107) from Day 0. Visual function of the study eye was assessed using the ETDRS protocol, which is a widely accepted international standard. A higher letter score represents better functioning"
Time Frame: 2 Years
Population: For those lost to follow-up, last observation carried forward
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
units on a scale | 72.5 [67.25 to 81.5] | 75.0 [69.0 to 80.0] | 75.0 [69.8 to 82.3]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events, ocular and non-ocular, in each of the study groups
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Participants
  Ocular Adverse Events : Blepharitis | 0 | 1 | 0
  Ocular Adverse Events : Blurred Vision/Vision Loss | 1 | 6 | 5
  Ocular Adverse Events : Cataract Progression | 1 | 5 | 7
  Ocular Adverse Events : Chalazion | 2 | 0 | 1
  Ocular Adverse Events : Conjunctivitis | 1 | 0 | 1
  Ocular Adverse Events : Conjunctival hemorrhage | 0 | 2 | 2
  Ocular Adverse Events : Corneal Abrasion | 0 | 0 | 1
  Ocular Adverse Events : Corneal Edema | 0 | 2 | 0
  Ocular Adverse Events : Diplopia | 0 | 0 | 1
  Ocular Adverse Events : Dysphotopsia | 0 | 1 | 0
  Ocular Adverse Events : Elevated IOP | 3 | 4 | 3
  Ocular Adverse Events : Epiretinal Membrane | 1 | 1 | 1
  Ocular Adverse Events : Eye discomfort/discharge | 6 | 9 | 15
  Ocular Adverse Events : Eyelid Swelling | 0 | 3 | 0
  Ocular Adverse Events : Glaucoma Progression | 0 | 1 | 1
  Ocular Adverse Events : Hollenhorst Plaque | 0 | 1 | 0
  Ocular Adverse Events : Macular Hole | 0 | 1 | 0
  Ocular Adverse Events : Optic Neuropathy | 1 | 2 | 0
  Ocular Adverse Events : Photophobia | 0 | 1 | 0
  Ocular Adverse Events : Pingueculum | 1 | 0 | 0
  Ocular Adverse Events : Secondary Cataract | 3 | 2 | 2
  Ocular Adverse Events : Vitreous floaters | 7 | 6 | 7
  Ocular Adverse Events : Punctate Keratitis | 2 | 3 | 6
  Ocular Adverse Events : Retinal Hemorrhage | 0 | 1 | 0
  Ocular Adverse Events : Vitreomacular Traction | 1 | 1 | 0
  Ocular Adverse Events : Vitreous Hemorrhage | 0 | 4 | 1
  Ocular Adverse Events : Vitritis | 0 | 1 | 0
  Ocular Adverse Events : Worsening Retinopathy | 1 | 2 | 2
  Nonocular AE: Acute Myocardial Infarction | 0 | 5 | 2
  Nonocular AE: Angina Pectoris | 0 | 0 | 5
  Nonocular AE: Arrhythmia | 2 | 1 | 3
  Nonocular AE: Cardiomyopathy | 0 | 1 | 0
  Nonocular AE: Congestive Heart Failure | 0 | 2 | 4
  Nonocular AE: Coronary Artery Disease | 0 | 2 | 2
  Nonocular AE: Pericardial Effusion | 0 | 0 | 1
  Nonocular AE: Peripheral Edema | 1 | 6 | 8
  Nonocular AE: Constipation | 0 | 2 | 2
  Nonocular AE: Diverticulitis | 1 | 1 | 0
  Nonocular AE: Diarrhea | 2 | 0 | 1
  Nonocular AE: Elevated liver enzymes | 1 | 0 | 0
  Nonocular AE: Nausea/emesis | 1 | 1 | 2
  Nonocular AE: Gallstones | 1 | 1 | 3
  Nonocular AE: Esophageal Reflux | 2 | 4 | 3
  Nonocular AE: Hemorrhoids | 1 | 1 | 0
  Nonocular AE: Incontinence | 1 | 0 | 0
  Nonocular AE: Poor dentition | 2 | 3 | 3
  Nonocular AE: Throat Irritation | 3 | 1 | 1
  Nonocular AE: Anemia | 1 | 4 | 7
  Nonocular AE: Hematoma | 1 | 0 | 0
  Nonocular AE: Thrombocytopenia | 0 | 0 | 1
  Nonocular AE: Allergy | 5 | 9 | 5
  Nonocular AE: Appendicitis | 1 | 0 | 0
  Nonocular AE: Epistaxis | 1 | 0 | 1
  Nonocular AE: Fever | 2 | 2 | 1
  Nonocular AE: Gastrointestinal infection | 1 | 3 | 4
  Nonocular AE: Parotitis | 0 | 0 | 1
  Nonocular AE: Skin Infection | 6 | 18 | 20
  Nonocular AE: Respiratory Infection | 12 | 22 | 14
  Nonocular AE: Sinusitis | 5 | 9 | 3
  Nonocular AE: Urinary Tract Infection | 4 | 2 | 1
  Nonocular AE: Elevated Creatinine | 0 | 0 | 2
  Nonocular AE: Fatigue | 3 | 1 | 0
  Nonocular AE: Graves disease | 1 | 0 | 0
  Nonocular AE: Hyperammonemia | 1 | 0 | 0
  Nonocular AE: Hypo/hyperglycemia | 7 | 12 | 14
  Nonocular AE: Hyperlipidemia | 5 | 4 | 6
  Nonocular AE: Hypo/hypercalcemia | 0 | 0 | 1
  Nonocular AE: Hypo/hyperkalemia | 0 | 1 | 5
  Nonocular AE: Hypothyroidism/nodule | 1 | 1 | 0
  Nonocular AE: Hyperparathyroidism | 0 | 0 | 1
  Nonocular AE: Hyperphosphatemia | 0 | 0 | 2
  Nonocular AE: Hyperuricemia | 0 | 0 | 1
  Nonocular AE: Testosterone deficiency | 2 | 1 | 0
  Nonocular AE: Vitamin D Deficiency | 1 | 3 | 2
  Nonocular AE: Weight Gain | 1 | 1 | 0
  Nonocular AE: Arthritis | 1 | 1 | 1
  Nonocular AE: Fractured Bone | 2 | 3 | 9
  Nonocular AE: Hernia | 0 | 0 | 1
  Nonocular AE: Musculoskeletal Pain | 12 | 16 | 18
  Nonocular AE: Osteoporosis | 0 | 0 | 1
  Nonocular AE: Skin burn | 2 | 2 | 1
  Nonocular AE: Colon Cancer | 1 | 3 | 1
  Nonocular AE: Lung Cancer | 1 | 0 | 1
  Nonocular AE: Prostate Cancer | 0 | 1 | 0
  Nonocular AE: Skin Cancer | 1 | 0 | 2
  Nonocular AE: Cranial Nerve Palsy | 0 | 0 | 2
  Nonocular AE: Cerebrovascular Accident | 0 | 0 | 3
  Nonocular AE: Decreased Hearing | 0 | 1 | 1
  Nonocular AE: Depression/Anxiety | 0 | 1 | 3
  Nonocular AE: Dizziness | 1 | 3 | 1
  Nonocular AE: Headache | 6 | 1 | 3
  Nonocular AE: Insomnia | 7 | 7 | 0
  Nonocular AE: Neuropathy | 1 | 0 | 1
  Nonocular AE: Paresthesia | 2 | 1 | 1
  Nonocular AE: Syncope/Presyncope | 1 | 2 | 2
  Nonocular AE: Seizure | 0 | 1 | 0
  Nonocular AE: Tinnitus | 0 | 1 | 1
  Nonocular AE: Transient Ischemic Attack | 0 | 0 | 1
  Nonocular AE: Kidney Stone | 1 | 2 | 1
  Nonocular AE: Renal Insufficiency | 1 | 1 | 6
  Nonocular AE: Acute Respiratory Failure | 1 | 1 | 1
  Nonocular AE: Cough | 2 | 5 | 5
  Nonocular AE: Dyspnea | 0 | 2 | 2
  Nonocular AE: Lung Nodule | 0 | 1 | 0
  Nonocular AE: Pneumonia | 2 | 4 | 3
  Nonocular AE: Pulmonary Embolism | 0 | 0 | 1
  Nonocular AE: Rhinorrhea | 0 | 0 | 1
  Nonocular AE: Sleep apnea | 0 | 0 | 1
  Nonocular AE: Orthostatic Hypotension | 0 | 1 | 0
  Nonocular AE: Peripheral Vascular Disease | 0 | 0 | 1
  Nonocular AE: Worsening Hypertension | 10 | 21 | 26

3. Secondary Outcome: Number of Intravitreal Injections
Description: Total number of intravitreal injections required during the first 12 months (week 46 - week 57) and the entire 24-month (week 92 - week 107) study period.
Time Frame: 2 years
Population: Multiple imputation model for eyes lost to follow-up prior to week 104 visit.
Measure: Median (Inter-Quartile Range); unit: Injections
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Injections | 25.0 [24.0 to 26.0] | 19.0 [13.8 to 24.0] | 17.0 [12.0 to 21.3]

4. Secondary Outcome: Number of Office Visits
Description: Total number of office visits and imaging studies performed during the first 12 months (week 46 - week 57) and the entire 24-month (week 92 - week 107) study period.
Time Frame: 2 years
Population: Multiple imputation model for eyes not reaching week 104 end-point visit.
Measure: Median (Inter-Quartile Range); unit: Visits
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Visits | 25.0 [24.0 to 26.0] | 19.0 [13.8 to 24.0] | 17.0 [12.0 to 21.3]

5. Secondary Outcome: Change in Retinal Thickness
Description: Mean change in central foveal thickness per SDOCT (Spectral Domain Optical Coherence Tomography) from randomization to 12 months (week46 - week 57) and randomization to 24 months (week 92 - week 107) study period.Change at month 24 reported.
Time Frame: 2 years
Population: For those not reaching week 104 end-point, last observation carried forward
Measure: Median (Inter-Quartile Range); unit: Microns
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Microns | 149 [75 to 234] | 151 [111 to 179] | 196 [85 to 266]

6. Secondary Outcome: Percentage of Eyes Gaining or Losing Vision
Description: Percentage of eyes gaining or losing 3 lines of vision or more and 1 line of vision at 24 months (week 92 - week 107) from Day 0.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Number analyzed (Eyes) | 30 | 60 | 60
Eyes
  1-line vision gainers | 13 | 28 | 32
  1-line vision losers | 5 | 1 | 3
  3-line vision gainers | 6 | 12 | 15
  3-line vision losers | 0 | 0 | 0

7. Secondary Outcome: Percentage of Eyes Which Progress to Proliferative Diabetic Retinopathy
Description: The percentage of eyes which show progression of proliferative diabetic retinopathy requiring panretinal photocoagulation and/or pars plana vitrectomy over the 24-month study period.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Number analyzed (Eyes) | 30 | 60 | 60
Eyes | 1 | 2 | 2

8. Secondary Outcome: Percentage of Eyes Able to Begin Extension Phase Prior to Week 104 End-point Visit.
Description: The percentage of eyes in the TREX (Treat and Extend) and GILA (Guided Laser) cohorts who are eligible to begin the extension phase prior to week 104 end-point visit.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Number analyzed (Eyes) | 30 | 60 | 60
Eyes | 0 | 49 | 55

9. Secondary Outcome: Percentage of Eyes With a Secondary or Tertiary Baseline Retinal Thickness
Description: For TREX and GILA Cohorts, the time to achieve a "Secondary or Tertiary Baseline" retinal thickness.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Monthly | TREX | GILA
Number analyzed (Participants) | 30 | 60 | 60
Number analyzed (Eyes) | 30 | 60 | 60
Eyes | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Monthly | TREX | GILA
All-Cause Mortality (participants affected / at risk) | 1/30 | 5/60 | 2/60
Serious Adverse Events (participants affected / at risk) | 11/30 | 30/60 | 46/60
Other Adverse Events (participants affected / at risk) | 30/30 | 60/60 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly (N=30) | TREX (N=60) | GILA (N=60)
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Vitreous Hemorrhage
Myocardial Infarction (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2) — Myocardial Infarction
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Angina Pectoris
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) — Cardiac Arrhythmia
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Cardiomyopathy
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4) — Congestive Heart Failure
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) — Coronary Artery Disease
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Pericardial Effusion
Gallstones (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Gallstones
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Hematoma
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Thrombocytopenia
Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Allergy
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Appendicitis
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Gastrointestinal Infection
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Parotitis
Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Respiratory Infection
Skin/Soft Tissue Infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) — Skin/Soft Tissue Infection
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Urinary Tract Infection
Elevated Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Elevated Creatinine
Hyperammonemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Hyperammonemia
Hypo/Hyperglycemia (Endocrine disorders) | 0 (0) | 2 (2) | 2 (2) — Hypo/Hyperglycemia
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Osteoarthritis
Fractured Bone (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) — Fractured Bone
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Musculoskeletal Pain
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) — Colon Cancer
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) — Lung Cancer
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Prostate Cancer
Cranial Nerve Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Cranial Nerve Palsy
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) — Cerebrovascular Accident
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — Syncope
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Transient Ischemic Attack
Urolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) — Urolithiasis
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) — Renal Failure
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) — Acute Respiratory Failure
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Dyspnea
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 3 (3) — Pneumonia
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Orthostatic Hypotension
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 6 (6) — Hypertension
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly (N=30) | TREX (N=60) | GILA (N=60)
Blurred Vision/Vision Loss (Eye disorders) | 1 (1) | 6 (6) | 5 (5) — Blurred Vision/Vision Loss
Cataract Progression (Eye disorders) | 1 (1) | 5 (5) | 7 (7) — Cataract Progression
Chalazion (Eye disorders) | 2 (2) | 0 (0) | 1 (1) — Chalazion
Elevated Intraocular Pressure (Eye disorders) | 3 (3) | 4 (4) | 3 (3) — Elevated Intraocular Pressure
Eye Discomfort/Discharge (Eye disorders) | 6 (6) | 9 (9) | 15 (15) — Eye Discomfort/Discharge
Eyelid Swelling (Eye disorders) | 0 (0) | 3 (3) | 0 (0) — Eyelid Swelling
Secondary Cataract (Eye disorders) | 3 (3) | 2 (2) | 2 (2) — Secondary Cataract
Vitreous Floaters (Eye disorders) | 7 (7) | 6 (6) | 7 (7) — Vitreous Floaters
Punctate Keratitis (Eye disorders) | 2 (2) | 3 (3) | 6 (6) — Punctate Keratitis
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 4 (4) | 1 (1) — Vitreous Hemorrhage
Myocardial Infarction (Cardiac disorders) | 0 (0) | 5 (5) | 2 (2) — Myocardial Infarction
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5) — Angina Pectoris
Cardiac Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3) — Cardiac Arrhythmia
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4) — Congestive Heart Failure
Peripheral Edema (Vascular disorders) | 1 (1) | 6 (6) | 8 (8) — Peripheral Edema
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) — Diarrhea
Gallstones (Hepatobiliary disorders) | 1 (1) | 1 (1) | 3 (3) — Gallstones
Esophageal Reflux (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) — Esophageal Reflux
Poor Dentition (General disorders) | 2 (2) | 3 (3) | 3 (3) — Poor Dentition
Throat Irritation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) — Throat Irritation
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 7 (7) — Anemia
Allergy (Immune system disorders) | 5 (5) | 9 (9) | 5 (5) — Allergy
Fever (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) — Fever
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) — Gastrointestinal Infection
Skin Infection (Infections and infestations) | 6 (6) | 18 (18) | 20 (20) — Skin Infection
Respiratory Infection (Infections and infestations) | 12 (12) | 22 (22) | 14 (14) — Respiratory Infection
Sinusitis (Infections and infestations) | 5 (5) | 9 (9) | 3 (3) — Sinusitis
Urinary Tract Infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) — Urinary Tract Infection
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0) — Fatigue
Hypo/Hyperglycemia (Endocrine disorders) | 7 (7) | 12 (12) | 14 (14) — Hypo/Hyperglycemia
Hyperlipidemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 6 (6) — Hyperlipidemia
Hypo/Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) — Hypo/Hyperkalemia
Testosterone Deficiency (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) — Testosterone Deficiency
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) — Vitamin D Deficiency
Fractured Bone (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 9 (9) — Fractured Bone
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 16 (16) | 18 (18) — Musculoskeletal Pain
Skin Burn (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) — Skin Burn
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 1 (1) — Colon Cancer
Depression/Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) — Depression/Anxiety
Dizziness (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 1 (1) — Dizziness
Headache (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 3 (3) — Headache
Insomnia (General disorders) | 7 (7) | 7 (7) | 0 (0) — Insomnia
Paresthesia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) — Paresthesia
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1) | 6 (6) — Renal Insufficiency
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 5 (5) — Cough
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) — Pneumonia
Hypertension (Vascular disorders) | 10 (10) | 21 (21) | 26 (26) — Hypertension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT01934556/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT01934556/ICF_001.pdf